CLINICAL TRIAL: NCT02955069
Title: An Open Label Phase II Study to Evaluate the Efficacy and Safety of PDR001 in Patients With Advanced or Metastatic, Well-differentiated, Non-functional Neuroendocrine Tumors of Pancreatic, Gastrointestinal (GI), or Thoracic Origin or Poorly-differentiated Gastroenteropancreatic Neuroendocrine Carcinoma (GEP-NEC), That Have Progressed on Prior Treatment.
Brief Title: Study of Efficacy and Safety of PDR001 in Patients With Advanced or Metastatic, Well-differentiated, Non-functional Neuroendocrine Tumors of Pancreatic, Gastrointestinal (GI), or Thoracic Origin or Poorly-differentiated Gastroenteropancreatic Neuroendocrine Carcinoma (GEP-NEC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPDR001E2201; 2016-002522-36 (EudraCT Number)
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Results first posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-03

CONDITIONS: Well-differentiated Non-functional NET of Thoracic Origin; Well-differentiated Non-functional NET of Gastrointestinal Origin; Well-differentiated Non-functional NET of Pancreatic Origin; Poorly-differentiated Gastroenteropancreatic Neuroendocrine Carcinoma
Keywords: Advanced or metastatic; NET; pNET; GI NET; thoracic NET; GEP-NEC
MeSH Terms: conditions — Neoplasm Metastasis; Neuroectodermal Tumors, Primitive | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PDR001 (Experimental): Subjects with advanced or metastatic, well-differentiated, NET of pancreatic, GI, or thoracic origin or poorly-differentiated GEP-NEC, that have progressed on prior treatment were treated with 400mg PDR001 administered via intravenous infusion once every 4 weeks.
  Interventions: Drug: PDR001

INTERVENTIONS:
Drug: PDR001 — PDR001 was administered at a dose of 400 mg via intravenous infusion once every 4 weeks (Q4W). PDR001 was administered on Day 1 of every cycle. Each cycle was 28 days.
  Other Names: Spartalizumab

SUMMARY:
This study aimed to investigate the efficacy and safety of PDR001 in patients with advanced or metastatic, well-differentiated, non-functional neuroendocrine tumors of pancreatic, gastrointestinal (GI), or thoracic origin or poorly-differentiated gastroenteropancreatic neuroendocrine carcinoma (GEP-NEC) that progressed on prior treatment.

DETAILED DESCRIPTION:
Two groups of adult patients with advanced (unresectable or metastatic) were included in this study:

* Well-differentiated (G1/2), non-functional, neuroendocrine tumor of GI, pancreatic or thoracic (lung/thymus) origin who have progressed on prior treatment
* Poorly-differentiated GEP-NEC who have progressed on or after one prior chemotherapy regimen.

The study was comprised of the following periods: screening, treatment, end of treatment (EOT), safety follow-up (30-Days, 60-Days, 90-Days, 120-Days, and 150-Days after the last dose of PDR001) and post-treatment efficacy follow-up. Subjects were treated with PDR001 as an infusion at a flat dose of 400 mg every 4 weeks (Q4W). Subjects were to continue study treatment beyond disease progression by RECIST 1.1 until disease progression as per irRECIST, as per BIRC, unacceptable toxicity, start of new antineoplastic therapy, withdrawal of consent, physician's decision, lost to follow-up, death, or study termination by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed, advanced (unresectable or metastatic):
* Well-differentiated (G1 or G2) based on local pathology report, non-functional neuroendocrine tumor of GI, pancreatic or thoracic (including lung and thymus) origin.
* Poorly-differentiated GEP-NEC based on local pathology report
* No active symptoms related to carcinoid syndrome during the last 3 months prior to start of study treatment.
* Patients must have been pretreated for advanced disease - the number of prior systemic therapy/regimen depended on which origin for NET and for GEP-NEC
* Tumor biopsy material must be provided for all patients for the purpose of biomarker analysis
* Radiological documentation of disease progression:
* Well-differentiated NET group: Disease progression while on/or after the last treatment, and this progression must have been observed within 6 months prior to start of study treatment (i.e. maximum of 24 weeks from documentation of progression until study entry). Disease must show evidence of radiological disease progression based on scans performed not more than 12 months apart.
* Poorly-differentiated GEP-NEC group: Disease progression while on or after prior treatment.

Exclusion Criteria:

* Well-differentiated grade 3 neuroendocrine tumors; poorly-differentiated neuroendocrine carcinoma of any origin (other than GEP-NEC); including NEC of unknown origin, adenocarcinoid, and goblet cell carcinoid
* Pretreatment with interferon as last treatment prior to start of study treatment.
* Prior treatment for study indication with:
* Antibodies or immunotherapy within 6 weeks before the first dose of study treatment.
* Peptide Radionuclide Receptor Therapy (PRRT) administered within 6 months of the first dose.
* Systemic antineoplastic therapy
* Tyrosine kinase inhibitors within 14 days or 5 half-lives, whichever is longer, before the first dose of study treatment.
* Prior Programmed Death-1 (PD-1) or Programmed Death-Ligand 1 (PD-L1) directed therapy.
* Cryoablation, radiofrequency ablation, or trans-arterial embolization of hepatic metastases
* History of severe hypersensitivity reactions to other monoclonal antibodies which in the opinion of the investigator may pose an increased risk of a serious infusion reaction.

Other inclusion/exclusion criteria might apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2020-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (33):
- United States (7):
  - City of Hope National Medical Center, Duarte, California
  - Rocky Mountain Cancer Centers SC-2, Denver, Colorado
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of TX MD Anderson Cancer Center, Houston, Texas
- Novartis Investigative Site, St Leonards, New South Wales, Australia
- Novartis Investigative Site, Vienna, Austria
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- France (3):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Toulouse
- Germany (4):
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marburg
- Italy (5):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Meldola, FC
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Napoli
- Japan (4):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Chuo Ku, Tokyo
- Novartis Investigative Site, Amsterdam, Netherlands
- Spain (2):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in 35 investigative sites in 12 countries from 14 Feb 2017 to 04 Apr 2018
Pre-assignment Details: A total of 149 participants were screened. Those participants who met the eligibility criteria entered the treatment period.
Groups:
- Well-differentiated NET: Subjects with advanced or metastatic, well-differentiated non-functional NET of GI, pancreatic or thoracic origin that progressed on or after prior available treatments.
- Poorly-differentiated GEP-NEC: Subjects with advanced or metastatic poorly-differentiated GEP-NEC that progressed on or after prior available treatments.
Period: Overall Study
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC
Started | 95 | 21
Full Analysis Set (FAS) (All subjects to whom study treatment was assigned and who received at least one dose of PDR001.) | 95 | 21
Safety Set (All subjects who received at least one dose of PDR001.) | 95 | 21
Pharmacokinetic Analysis Set (PAS) (All subjects who provide at least one evaluable PDR001 pharmacokinetic (PK) concentration.) | 94 | 18
Immunogenicity (IG) Prevalence Set (All subjects in the FAS with a baseline or at least one post-baseline IG sample.) | 94 | 21
IG Incidence Set (All subjects in the IG prevalence set with a baseline and at least one post-baseline IG sample.) | 84 | 17
Completed | 0 | 0
Not Completed | 95 | 21
Not completed — Adverse Event | 7 | 2
Not completed — Death | 7 | 3
Not completed — Physician Decision | 10 | 2
Not completed — Progressive disease | 64 | 13
Not completed — Study terminated by sponsor | 4 | 0
Not completed — Subject/Guardian decision | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC | Total
Number analyzed (Participants) | 95 | 21 | 116
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.4 (11.21) | 57.4 (8.56) | 59.0 (10.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 4 | 47
  Male | 52 | 17 | 69
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 59 | 16 | 75
  Black | 4 | 0 | 4
  Asian | 7 | 3 | 10
  Native American | 1 | 0 | 1
  Black or African American | 2 | 0 | 2
  White | 15 | 1 | 16
  Unknown | 3 | 1 | 4
  Other | 3 | 0 | 3
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) by RECIST 1.1 and as Per Blinded Independent Central Review (BIRC).
Description: ORR is defined as the proportion of patients with best overall response (BOR) of complete response (CR) or partial response (PR), according to BIRC radiological assessment by RECIST 1.1.
  CR: disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
  PR: at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From baseline up to approximately 1.5 years
Population: The FAS comprised of all subjects to whom study treatment had been assigned and who received at least one dose of PDR001 (including incomplete infusion).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC
Number analyzed (Participants) | 95 | 21
Percentage of participants | 7.4 [3.0 to 14.6] | 4.8 [0.1 to 23.8]

2. Secondary Outcome: Duration of Response (DOR) by RECIST 1.1 and as Per BIRC
Description: DOR is defined as the time between the date of first documented response (CR or PR) and the date of first documented disease progression by RECIST 1.1 and as per BIRC or death due to underlying cancer. For DOR analysis, participants continuing without progression or death due to underlying cancer were censored at the date of their last adequate tumor assessment. An adequate tumour assessment is a tumour assessment with an overall response other than unknown.
  CR: disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
  PR: at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From the date of first documented response (CR or PR) until the first documented disease progression or death, whichever comes first, assessed up to approximately 1.5 years
Population: Participants in the FAS with confirmed CR or PR
Measure: Median (Full Range); unit: Days
Groups:
- Poorly Differentiated GEP-NEC: Subjects with advanced or metastatic poorly-differentiated GEP-NEC that progressed on or after prior available treatments.
Arm/Group | Well-differentiated NET | Poorly Differentiated GEP-NEC
Number analyzed (Participants) | 7 | 1
Days | 250 [49 to 288] | 270 [270 to 270]

3. Secondary Outcome: Disease Control Rate by RECIST 1.1 and as Per BIRC
Description: Disease control rate is defined as the proportion of patients with best overall response of CR, PR or stable disease (SD) according to RECIST 1.1 criteria and as per BIRC.
  CR: disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
  PR: at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  SD: neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: From baseline up to approximately 1.5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC
Number analyzed (Participants) | 95 | 21
Percentage of participants | 64.2 [53.7 to 73.8] | 19.0 [5.4 to 41.9]

4. Secondary Outcome: Time to Response (TTR) by RECIST 1.1 and as Per BIRC
Description: TTR is defined as the time from the date of start of treatment to the first documented response of either CR or PR, which must be subsequently confirmed. TTR was evaluated according to RECIST 1.1 and as per BIRC.
  CR: disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
  PR: at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From baseline to the first documented response, assessed up to approximately 1.5 years
Population: Participants in the FAS with confirmed CR or PR.
Measure: Median (Full Range); unit: Days
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC
Number analyzed (Participants) | 7 | 1
Days | 110 [52 to 218] | 53 [53 to 53]

5. Secondary Outcome: Progression-free Survival (PFS) by RECIST 1.1 and as Per BIRC
Description: PFS is defined as the time from the date of first dose to the date of the first documented radiological progression or death due to any cause. PFS was evaluated according to RECIST 1.1 and as per BIRC. For participants who had not progressed or died at the analysis cut-off date, PFS was censored at the date of the last adequate tumor evaluation date. An adequate tumour assessment is a tumour assessment with an overall response other than unknown.
Time Frame: From baseline until the date of the first documented radiological progression or death due to any cause, whichever comes first, assessed up to approximately 1.5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC
Number analyzed (Participants) | 95 | 21
Months | 3.8 [3.6 to 5.5] | 1.8 [1.5 to 2.0]

6. Secondary Outcome: Immune Related Overall Response Rate (irORR) by irRECIST and as Per BIRC
Description: irORR is the proportion of patients with a best overall response of immune related Complete Response (irCR) or immune related partial response (irPR), according to BIRC assessment by irRECIST.
  irCR: Complete disappearance of all measurable and non-measurable lesions. In addition, any pathological lymph nodes must have a reduction in short axis to < 10 mm.
  irPR: At least 30% decrease in the total measurable tumor burden (TMTB) compared to baseline and not qualifying for irCR or immune related progressive disease (irPD).
Time Frame: From baseline up to approximately 1.5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC
Number analyzed (Participants) | 95 | 21
Percentage of participants | 7.4 [3.0 to 14.6] | 4.8 [0.1 to 23.8]

7. Secondary Outcome: Immune Related Duration of Response (irDoR) by irRECIST and as Per BIRC.
Description: irDOR is defined as the time from first documentation of irCR or irPR until the time of first documentation of progression per irRECIST based on BIRC assessment. Participants continuing without progression or death due to underlying cancer were censored at the date of their last adequate tumor assessment. An adequate tumour assessment is a tumour assessment with an overall response other than unknown for irRECIST.
  irCR: Complete disappearance of all measurable and non-measurable lesions. In addition, any pathological lymph nodes must have a reduction in short axis to < 10 mm.
  irPR: At least 30% decrease in the TMTB compared to baseline and not qualifying for irPD or irCR
Time Frame: From the date of first documented confirmed response (irCR or irPR) until the first documented progression, assessed up to approximately 1.5 years
Population: Participants in the FAS with confirmed irCR or irPR
Measure: Median (Full Range); unit: Days
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC
Number analyzed (Participants) | 7 | 1
Days | 228 [49 to 288] | 270 [270 to 270]

8. Secondary Outcome: Immune Related Time to Response (irTTR) by irRECIST and as Per BIRC
Description: irTTR is defined as the time between date of start of treatment until first documented response (confirmed irCR or irPR) by irRECIST and as per BIRC.
  irCR: Complete disappearance of all measurable and non-measurable lesions. In addition, any pathological lymph nodes must have a reduction in short axis to < 10 mm.
  irPR: At least 30% decrease in the TMTB compared to baseline and not qualifying for irPD or irCR.
Time Frame: From baseline to the first documented response, assessed up to approximately 1.5 years
Population: Participants in the FAS with confirmed irCR or irPR
Measure: Median (Full Range); unit: Days
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC
Number analyzed (Participants) | 7 | 1
Days | 110 [52 to 218] | 53 [53 to 53]

9. Secondary Outcome: Immune Related Disease Control Rate (irDCR) by irRECIST and as Per BIRC
Description: irDCR is defined as the proportion of patients with a best overall response of irCR or irPR or immune related stable disease (irSD) according to irRECIST and as per BIRC.
  irCR: Complete disappearance of all measurable and non-measurable lesions. In addition, any pathological lymph nodes must have a reduction in short axis to < 10 mm.
  irPR: At least 30% decrease in the TMTB compared to baseline and not qualifying for irPD or irCR.
  irSD: Neither a sufficient shrinkage to qualify for irPR or irCR, nor an increase in lesions, or a clear and unequivocal progression of existing nontarget or new non-measurable lesions that would qualify for irPD.
Time Frame: From baseline up to approximately 1.5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC
Number analyzed (Participants) | 95 | 21
Percentage of participants | 66.3 [55.9 to 75.7] | 19.0 [5.4 to 41.9]

10. Secondary Outcome: Immune Related Progression Free Survival (irPFS) by irRECIST and as Per BIRC
Description: irPFS is defined as the time from date of start of treatment to the date of event defined as the first documented assessment of immune related progression that is confirmed or death due to any cause. If a patient has not had an event, immune related progression-free survival was censored at the date of last adequate tumor assessment. An adequate tumor assessment is a tumor assessment with overall response other than unknown for irRECIST.
Time Frame: From baseline until the date of the first documented immune related progression or death due to any cause, whichever comes first, assessed up to approximately 1.5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC
Number analyzed (Participants) | 95 | 21
Months | 3.8 [3.6 to 5.5] | 1.8 [1.5 to 2.0]

11. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the start of treatment date to the date of death, due to any cause. If a patient was not known to have died, then OS was censored at the latest date the patient was known to be alive.
Time Frame: From baseline until death due to any cause, assessed up to approx. 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC
Number analyzed (Participants) | 95 | 21
Months | 23.4 [19.2 to NA] — NA: Upper limit was not evaluable | 6.8 [4.0 to 8.6]

12. Secondary Outcome: Changes From Baseline in Chromogranin A (CgA) Levels
Description: Blood samples were collected for assessment of CgA level. Change from Baseline at a particular visit was calculated as the CgA level at that visit minus Baseline.
Time Frame: Baseline, day 1 of each cycle from Cycle 2 to end of treatment, assessed up to approx. 1.5 years. Cycle=28 days.
Population: The FAS comprised of all subjects to whom study treatment had been assigned and who received at least one dose of PDR001 (including incomplete infusion). Number analyzed signified number of participants with available data for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: microgram/liter (ug/L)
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC
Number analyzed (Participants) | 95 | 21
microgram/liter (ug/L)
  Cycle 2 Day 1: number analyzed (Participants) | 87 | 14
  Cycle 2 Day 1 | 874.6 (6694.64) | 6466.9 (23760.13)
  Cycle 3 Day 1: number analyzed (Participants) | 77 | 8
  Cycle 3 Day 1 | -1811.7 (21413.11) | 706.5 (2294.87)
  Cycle 4 Day 1: number analyzed (Participants) | 69 | 6
  Cycle 4 Day 1 | 579.9 (13437.06) | 1544.5 (2712.23)
  Cycle 5 Day 1: number analyzed (Participants) | 53 | 5
  Cycle 5 Day 1 | 598.2 (11724.93) | 1306.6 (3125.84)
  Cycle 6 Day 1: number analyzed (Participants) | 47 | 3
  Cycle 6 Day 1 | 1337.6 (7106.32) | 4531.7 (8694.65)
  Cycle 7 Day 1: number analyzed (Participants) | 41 | 2
  Cycle 7 Day 1 | -564.5 (12643.71) | 11089.5 (17551.10)
  Cycle 8 Day 1: number analyzed (Participants) | 29 | 2
  Cycle 8 Day 1 | 3726.0 (18813.63) | 9103.5 (14759.44)
  Cycle 9 Day 1: number analyzed (Participants) | 27 | 1
  Cycle 9 Day 1 | 22522.2 (94054.85) | -1342.0 (NA) — NA: Not evaluable due to low number of participants analyzed
  Cycle 10 Day 1: number analyzed (Participants) | 26 | 1
  Cycle 10 Day 1 | 54301.5 (250229.27) | -1376.0 (NA) — NA: Not evaluable due to low number of participants analyzed
  Cycle 11 Day 1: number analyzed (Participants) | 21 | 1
  Cycle 11 Day 1 | 84634.7 (344244.60) | -1393.0 (NA) — NA: Not evaluable due to low number of participants analyzed
  Cycle 12 Day 1: number analyzed (Participants) | 18 | 1
  Cycle 12 Day 1 | 8177.6 (36820.47) | -1362.0 (NA) — NA: Not evaluable due to low number of participants analyzed
  Cycle 13 Day 1: number analyzed (Participants) | 16 | 1
  Cycle 13 Day 1 | -379.8 (1509.95) | -1377.0 (NA) — NA: Not evaluable due to low number of participants analyzed
  Cycle 14 Day 1: number analyzed (Participants) | 15 | 0
  Cycle 14 Day 1 | 398.3 (1866.56) |
  Cycle 15 Day 1: number analyzed (Participants) | 12 | 0
  Cycle 15 Day 1 | 13.1 (1120.60) |
  Cycle 16 Day 1: number analyzed (Participants) | 4 | 0
  Cycle 16 Day 1 | -81.0 (1583.99) |
  Cycle 17 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 17 Day 1 | -176.0 (NA) — NA: Not evaluable due to low number of participants analyzed |
  Cycle 18 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 18 Day 1 | 42.0 (NA) — NA: Not evaluable due to low number of participants analyzed |
  End of treatment: number analyzed (Participants) | 34 | 7
  End of treatment | 30115.3 (131958.16) | 3899.6 (7991.40)

13. Secondary Outcome: Change From Baseline in Neuron Specific Enolase (NSE) Levels
Description: Blood samples were collected for assessment of NSE level. Change from Baseline at a particular visit was calculated as the NSE level at that visit minus Baseline.
Time Frame: Baseline, day 1 of each cycle from Cycle 2 to end of treatment, assessed up to approx. 1.5 years. Cycle= 28days
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: microgram/liter (ug/L)
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC
Number analyzed (Participants) | 95 | 21
microgram/liter (ug/L)
  Cycle 2 Day 1: number analyzed (Participants) | 81 | 13
  Cycle 2 Day 1 | 0.8 (29.71) | 27.9 (40.77)
  Cycle 3 Day 1: number analyzed (Participants) | 73 | 7
  Cycle 3 Day 1 | 2.5 (29.33) | 32.6 (56.87)
  Cycle 4 Day 1: number analyzed (Participants) | 66 | 2
  Cycle 4 Day 1 | -0.1 (14.98) | 21.9 (21.64)
  Cycle 5 Day 1: number analyzed (Participants) | 48 | 4
  Cycle 5 Day 1 | 4.8 (30.34) | 31.8 (56.39)
  Cycle 6 Day 1: number analyzed (Participants) | 43 | 2
  Cycle 6 Day 1 | -3.6 (19.18) | 151.6 (204.21)
  Cycle 7 Day 1: number analyzed (Participants) | 41 | 2
  Cycle 7 Day 1 | 7.6 (39.44) | -3.0 (17.75)
  Cycle 8 Day 1: number analyzed (Participants) | 25 | 1
  Cycle 8 Day 1 | 1.0 (22.19) | 40.4 (NA) — NA: Not evaluable due to low number of participants analyzed
  Cycle 9 Day 1: number analyzed (Participants) | 25 | 1
  Cycle 9 Day 1 | 2.6 (8.64) | -12.7 (NA) — NA: Not evaluable due to low number of participants analyzed
  Cycle 10 Day 1: number analyzed (Participants) | 21 | 1
  Cycle 10 Day 1 | 10.3 (33.74) | -15.0 (NA) — NA: Not evaluable due to low number of participants analyzed
  Cycle 11 Day 1: number analyzed (Participants) | 18 | 0
  Cycle 11 Day 1 | 2.3 (8.89) |
  Cycle 12 Day 1: number analyzed (Participants) | 17 | 1
  Cycle 12 Day 1 | -2.4 (23.04) | -12.3 (NA) — NA: Not evaluable due to low number of participants analyzed
  Cycle 13 Day 1: number analyzed (Participants) | 14 | 1
  Cycle 13 Day 1 | -3.9 (24.22) | -17.8 (NA) — NA: Not evaluable due to low number of participants analyzed
  Cycle 14 Day 1: number analyzed (Participants) | 15 | 0
  Cycle 14 Day 1 | -4.5 (22.71) |
  Cycle 15 Day 1: number analyzed (Participants) | 11 | 0
  Cycle 15 Day 1 | -3.4 (29.73) |
  Cycle 16 Day 1: number analyzed (Participants) | 3 | 0
  Cycle 16 Day 1 | 26.5 (35.38) |
  Cycle 17 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 17 Day 1 | 15.1 (NA) — NA: Not evaluable due to low number of participants analyzed |
  Cycle 18 Day 1: number analyzed (Participants) | 1 | 0
  Cycle 18 Day 1 | 13.8 (NA) — NA: Not evaluable due to low number of participants analyzed |
  End of treatment: number analyzed (Participants) | 33 | 7
  End of treatment | 47.7 (136.78) | 44.3 (66.73)

14. Secondary Outcome: PDR001 Plasma Concentration
Description: Blood samples will be taken to evaluate the pharmacokinetics by assessing plasma concentration of PDR001 at selected time points
Time Frame: Cycle(C)1 Day(D)1 pre-dose and 30min post-infusion,C2D1 Pre-dose,C3D1 Pre-dose and 30min post-infusion,D1 pre-dose from C4 to C13, assessed up to approx. 1.5 years.Cycle=28 days
Population: The PAS comprised of all subjects who provide at least one evaluable PDR001 PK concentration. Number analyzed signified number of participants with available data for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: nanogram/mililiter (ng/mL)
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC
Number analyzed (Participants) | 94 | 18
nanogram/mililiter (ng/mL)
  Cycle 1 Day 1 pre-dose: number analyzed (Participants) | 89 | 17
  Cycle 1 Day 1 pre-dose | 0 (0) | 0 (0)
  Cycle 1 Day 1 30 min post-dose: number analyzed (Participants) | 87 | 14
  Cycle 1 Day 1 30 min post-dose | 106 (32.9) | 100 (52.2)
  Cycle 2 Day 1 Pre-dose: number analyzed (Participants) | 85 | 14
  Cycle 2 Day 1 Pre-dose | 26.8 (9.76) | 25.8 (9.30)
  Cycle 3 Day 1 pre-dose: number analyzed (Participants) | 72 | 9
  Cycle 3 Day 1 pre-dose | 43.7 (18.9) | 42.3 (19.6)
  Cycle 3 Day 1 30 min post-dose: number analyzed (Participants) | 73 | 9
  Cycle 3 Day 1 30 min post-dose | 140 (46.7) | 142 (44.3)
  Cycle 4 Day 1 pre-dose: number analyzed (Participants) | 64 | 4
  Cycle 4 Day 1 pre-dose | 52.8 (25.1) | 40.7 (17.2)
  Cycle 5 Day 1 pre-dose: number analyzed (Participants) | 49 | 4
  Cycle 5 Day 1 pre-dose | 52.0 (32.3) | 41.8 (8.88)
  Cycle 6 Day 1 pre-dose: number analyzed (Participants) | 42 | 1
  Cycle 6 Day 1 pre-dose | 58.2 (31.6) | 49.9 (NA) — NA: Not evaluable due to low number of participants analyzed
  Cycle 7 Day 1 pre-dose: number analyzed (Participants) | 36 | 2
  Cycle 7 Day 1 pre-dose | 64.3 (37.6) | 66.9 (30.1)
  Cycle 8 Day 1 pre-dose: number analyzed (Participants) | 28 | 2
  Cycle 8 Day 1 pre-dose | 59.6 (38.2) | 64.7 (31.4)
  Cycle 9 Day 1 pre-dose: number analyzed (Participants) | 23 | 1
  Cycle 9 Day 1 pre-dose | 65.1 (38.1) | 93.7 (NA) — NA: Not evaluable due to low number of participants analyzed
  Cycle 10 Day 1 pre-dose: number analyzed (Participants) | 25 | 0
  Cycle 10 Day 1 pre-dose | 70.2 (40.2) |
  Cycle 11 Day 1 pre-dose: number analyzed (Participants) | 19 | 1
  Cycle 11 Day 1 pre-dose | 69.2 (39.1) | 99.0 (NA) — NA: Not evaluable due to low number of participants analyzed
  Cycle 12 Day 1 pre-dose: number analyzed (Participants) | 14 | 1
  Cycle 12 Day 1 pre-dose | 71.7 (38.1) | 111 (NA) — NA: Not evaluable due to low number of participants analyzed
  Cycle 13 Day 1 pre-dose: number analyzed (Participants) | 13 | 0
  Cycle 13 Day 1 pre-dose | 91.8 (46.0) |

15. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status/Quality of Life Score
Description: The EORTC QLQ-C30 is a patient completed 30 item questionnaire that is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, six single items and a global health status/QoL scale. Global health status/QoL response options are 1 to 4. Scores were averaged and transformed to 0 to 100. Higher scores indicate better functioning.
  Change from Baseline was calculated by subtracting Baseline value from the selected visit value. A positive change from Baseline indicates improvement.
Time Frame: Baseline, every 8 weeks from Cycle 3 Day 1 for the first 13 cycles and every 12 weeks from Cycle 13 Day 1 thereafter and end of treatment, assessed up to approx. 1.5 years. Cycle=28 days
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC
Number analyzed (Participants) | 95 | 21
score on a scale
  Cycle 3 Day 1: number analyzed (Participants) | 67 | 9
  Cycle 3 Day 1 | -1.00 (19.491) | -11.11 (27.003)
  Cycle 5 Day 1: number analyzed (Participants) | 48 | 4
  Cycle 5 Day 1 | -1.91 (27.838) | -4.17 (17.347)
  Cycle 7 Day 1: number analyzed (Participants) | 34 | 2
  Cycle 7 Day 1 | 1.96 (29.945) | 25.00 (35.355)
  Cycle 9 Day 1: number analyzed (Participants) | 25 | 1
  Cycle 9 Day 1 | 1.67 (31.823) | 33.33 (NA) — NA: Not evaluable due to low number of participants analyzed
  Cycle 11 Day 1: number analyzed (Participants) | 21 | 0
  Cycle 11 Day 1 | -1.19 (28.048) |
  Cycle 13 Day 1: number analyzed (Participants) | 17 | 1
  Cycle 13 Day 1 | 1.96 (27.088) | 41.67 (NA) — NA: Not evaluable due to low number of participants analyzed
  Cycle 16 Day 1: number analyzed (Participants) | 3 | 0
  Cycle 16 Day 1 | -16.67 (16.667) |
  End of Treatment: number analyzed (Participants) | 40 | 8
  End of Treatment | -6.46 (23.607) | -22.92 (23.465)

16. Secondary Outcome: Change From Baseline in EQ-5D-5L Index Score
Description: The EQ-5D-5L descriptive system provides a profile of the participant's health state in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each of these dimensions, the participant self-assigned a score: from 1 (no problems) to 5 (extreme problems). The 5 digit health states obtained for each dimension was converted into a single mean index value based on the EQ-5D crosswalk value set for the UK using the time trade-off method. This index ranges from -0.594 (worst health) to 1.0 (best health). Change from Baseline was calculated by subtracting Baseline value from the selected visit value. A positive change from baseline indicates improvement.
Time Frame: Baseline, every 8 weeks from Cycle 3 Day 1 for the first 13 cycles and every 12 weeks from Cycle 13 Day 1 thereafter, and end of treatment, assessed up to approx.1.5 year. Cycle=28 days
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC
Number analyzed (Participants) | 95 | 21
score on a scale
  Cycle 3 Day 1: number analyzed (Participants) | 66 | 8
  Cycle 3 Day 1 | 0.03 (0.169) | -0.09 (0.157)
  Cycle 5 Day 1: number analyzed (Participants) | 48 | 4
  Cycle 5 Day 1 | -0.02 (0.247) | 0.02 (0.111)
  Cycle 7 Day 1: number analyzed (Participants) | 33 | 2
  Cycle 7 Day 1 | -0.04 (0.241) | 0.16 (0.135)
  Cycle 9 Day 1: number analyzed (Participants) | 25 | 1
  Cycle 9 Day 1 | 0.02 (0.247) | 0.02 (NA) — NA: Not evaluable due to low number of participants analyzed
  Cycle 11 Day 1: number analyzed (Participants) | 21 | 0
  Cycle 11 Day 1 | 0.02 (0.262) |
  Cycle 13 Day 1: number analyzed (Participants) | 16 | 1
  Cycle 13 Day 1 | -0.03 (0.299) | 0.03 (NA) — NA: Not evaluable due to low number of participants analyzed
  Cycle 16 Day 1: number analyzed (Participants) | 3 | 0
  Cycle 16 Day 1 | -0.17 (0.085) |
  End of treatment: number analyzed (Participants) | 40 | 8
  End of treatment | -0.10 (0.209) | -0.30 (0.263)

17. Secondary Outcome: PDR001 Anti-drug Antibodies (ADA) Prevalence at Baseline
Description: ADA prevalence at baseline was calculated as the proportion of participants who had an ADA positive result at baseline
Time Frame: Baseline
Population: Participants in the Immunogenicity (IG) set with at least one determinant sample (sample that is neither ADA-inconclusive nor unevaluable) at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC
Number analyzed (Participants) | 88 | 17
Participants | 1 | 0

18. Secondary Outcome: PDR001 ADA Incidence On-treatment
Description: ADA incidence on treatment was calculated as the proportion of participants who were treatment-induced ADA positive (post-baseline ADA positive with ADA-negative sample at baseline) and treatment-boosted ADA positive (post-baseline ADA positive with titer that is at least the fold titer change greater than the ADA-positive baseline titer)
Time Frame: Cycle(C)1 Day(D)1 pre-dose and 30min post-infusion,C2D1 Pre-dose,C3D1 Pre-dose and 30min post-infusion,D1 pre-dose from C4 to C13 and every 6 cycles until C25, and end of treatment, assessed up to approx. 1.5 years. Cycle=28 days
Population: The IG incidence set comprised of all subjects in the IG prevalence set with a determinant baseline IG sample and at least one determinant post-baseline IG sample. Determinant sample: sample that is neither ADA-inconclusive nor unevaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC
Number analyzed (Participants) | 84 | 17
Participants | 10 | 2

19. Post Hoc Outcome: All Collected Deaths
Description: Deaths on-treatment are collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of approximately 3 years.
  Total Deaths are collected from first dose of study treatment until end of post-treatment efficacy or survival follow, up to maximum duration of approximately 3 years.
Time Frame: up to 3 years
Population: The Safety Set comprised all subjects who received at least one dose of PDR001
Measure: Number; unit: Participants
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC
Number analyzed (Participants) | 95 | 21
Participants
  Total Deaths | 47 | 16
  Deaths on-treatment | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of approximately 3 years.
Description: Any sign or symptom that occurs during the study treatment plus 30 days post treatment
Groups:
- All Subjects: All subjects
Arm/Group | Well-differentiated NET | Poorly-differentiated GEP-NEC | All Subjects
All-Cause Mortality (participants affected / at risk) | 1/95 | 1/21 | 2/116
Serious Adverse Events (participants affected / at risk) | 29/95 | 6/21 | 35/116
Other Adverse Events (participants affected / at risk) | 86/95 | 18/21 | 104/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Well-differentiated NET (N=95) | Poorly-differentiated GEP-NEC (N=21) | All Subjects (N=116)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Torsade de pointes (Cardiac disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 1 | 7
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2
Generalised oedema (General disorders) | 1 | 0 | 1
Malaise (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 3 | 0 | 3
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 1 | 1
Insulin autoimmune syndrome (Immune system disorders) | 1 | 0 | 1
Candida infection (Infections and infestations) | 1 | 0 | 1
Febrile infection (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 1
Systemic infection (Infections and infestations) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 1
Device occlusion (Product Issues) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Well-differentiated NET (N=95) | Poorly-differentiated GEP-NEC (N=21) | All Subjects (N=116)
Anaemia (Blood and lymphatic system disorders) | 18 | 3 | 21
Hypothyroidism (Endocrine disorders) | 7 | 0 | 7
Abdominal distension (Gastrointestinal disorders) | 5 | 2 | 7
Abdominal pain (Gastrointestinal disorders) | 17 | 1 | 18
Abdominal pain upper (Gastrointestinal disorders) | 7 | 0 | 7
Constipation (Gastrointestinal disorders) | 19 | 3 | 22
Diarrhoea (Gastrointestinal disorders) | 26 | 4 | 30
Dry mouth (Gastrointestinal disorders) | 5 | 0 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2 | 4
Nausea (Gastrointestinal disorders) | 20 | 5 | 25
Vomiting (Gastrointestinal disorders) | 11 | 3 | 14
Asthenia (General disorders) | 12 | 2 | 14
Fatigue (General disorders) | 36 | 3 | 39
Oedema peripheral (General disorders) | 14 | 3 | 17
Pain (General disorders) | 2 | 2 | 4
Pyrexia (General disorders) | 24 | 2 | 26
Infection (Infections and infestations) | 0 | 2 | 2
Alanine aminotransferase increased (Investigations) | 3 | 3 | 6
Amylase increased (Investigations) | 5 | 1 | 6
Aspartate aminotransferase increased (Investigations) | 1 | 4 | 5
Blood alkaline phosphatase increased (Investigations) | 3 | 3 | 6
Gamma-glutamyltransferase increased (Investigations) | 6 | 3 | 9
Lipase increased (Investigations) | 6 | 1 | 7
Weight decreased (Investigations) | 9 | 1 | 10
Weight increased (Investigations) | 4 | 2 | 6
Decreased appetite (Metabolism and nutrition disorders) | 15 | 3 | 18
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 1 | 8
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 | 0 | 8
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 0 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 0 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 2 | 14
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 0 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 0 | 7
Headache (Nervous system disorders) | 8 | 1 | 9
Anxiety (Psychiatric disorders) | 7 | 0 | 7
Insomnia (Psychiatric disorders) | 3 | 2 | 5
Proteinuria (Renal and urinary disorders) | 6 | 1 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 2 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 15
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 1 | 9
Rash (Skin and subcutaneous tissue disorders) | 10 | 2 | 12
Hypertension (Vascular disorders) | 12 | 0 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT02955069/SAP_000.pdf
  • Study Protocol (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT02955069/Prot_001.pdf